CLINICAL TRIAL: NCT00405509
Title: The Natural History of Viral Upper Respiratory Infections in Children Aged 6 to <14 Years
Brief Title: The Natural History of Viral Upper Respiratory Infections in Children Aged 6 to Less Than 14 Years
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Collaborators: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Deborah Gentile, Director of Research, Allergy and Asthma Institute, West Penn Allegheny Health System
Other Study IDs: RC#4065
Record Dates: First submitted 2006-11-28; First posted 2006-11-30 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Upper Respiratory Infection; Common Cold
Keywords: Upper Respiratory Infection; Common Cold
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal brushing for genotyping

GROUPS / COHORTS (2):
- Confirmed respiratory virus
- Unconfirmed respiratory infection

SUMMARY:
This study examines the cold processes of children aged 6 to less than 14. Children will be seen by the study staff 6 days in a row during the course of their naturally-acquired colds. Nasal secretions will be examined for chemicals that the body creates during a cold. Skin cells will be collected by brushing the inside of the child's cheek with a small brush. The cells will be examined for genes that may hold control the creation of these chemicals.

DETAILED DESCRIPTION:
Leukotrienes are chemicals that are naturally made by your body. Leukotrienes are increased in the bodies of adults and children with asthma and allergies and cause some of the symptoms of these diseases. Leukotrienes are increased in the bodies of adults who have common colds and are believed to cause some of the symptoms of the common cold. It is not known if increases in leukotrienes are related to the symptoms of the common cold in children. There are also genes that may control levels of leukotrienes and other chemicals in your body during the common cold. If you enroll your child in this study, he/she will be tested for allergies and for genes that may control the levels of leukotrienes and other chemicals.

STUDY DESIGN:

There will be 40 subjects enrolled into the study between the ages of 6 to < 14 years of age. However, approximately 80 participants may have to sign the consent form and undergo screening activities in order enroll these 40 subjects. The study will last approximately 1 month and will require you and your child to return to our clinic approximately 7 times over the study duration. You and your child will be required to return to our clinic six days in a row for testing.

Testing will include skin testing for allergies, nasal secretion collection, and skin cell collection.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to < 14 years of age.
* Common cold symptoms for less than 24 hours.
* At least 2 of the following 8 symptoms: cough, headache, hoarseness, muscle ache, nasal drainage, nasal congestion, scratchy throat, and sneezing.

Exclusion Criteria:

* Investigational medication in past 30 days.
* History of persistent asthma or other chronic diseases.
* Patients with nasal ulcers within the past 1 month, nasal surgery within the past 6 months, nasal trauma within the past 2 months or presence of nasal polyps or nasal deformities causing significant nasal obstruction.
* Patients with evidence of significant nasal septal deviation.
* Patients with a positive rapid antigen test for streptococcal infection.
* Common cold symptoms for more than 24 hours.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male and Female subjects ages 6 to under 14 years with common cold symptoms of less than 24 hours in duration.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gentile, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from private practice pediatric and family practice offices. Some subjects were recruited via Institutional Review Board (IRB)-approved advertisement.
Groups:
- Confirmed Respiratory Infection: respiratory infection virus type confirmed by assay
- Unconfirmed Respiratory Infection: participants who were not positive for any of the tested viruses and thus viral infection type could not be confirmed
Period: Overall Study
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Started | 11 | 22
Completed | 11 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Confirmed Respiratory Infection: participants who had the type of viral infection confirmed by assay
- Total: Total of all reporting groups
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection | Total
Number analyzed (Participants) | 11 | 22 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 22 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 9.0 (2.2) | 9.6 (2.3) | 9.4 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 15 | 19
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 11 | 22 | 33

OUTCOME MEASURES:

1. Primary Outcome: Local Leukotriene Levels
Description: nasal secretions were collected once a day for the first six days of the respiratory infection and on day 30 then measured for leukotriene levels
Time Frame: once a day for 6 days and on day 30
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Number analyzed (Participants) | 11 | 22
pg/ml
  Day 1 | 440 (70.34) | 368 (56.54)
  Day 2 | 440 (48.78) | 619 (103.21)
  Day 3 | 676 (136.87) | 368 (75.94)
  Day 4 | 992 (306.84) | 300 (50.51)
  Day 5 | 737 (310.34) | 530 (98.35)
  Day 6 | 624 (145.6) | 753 (185.8)
  Day 30 | 479 (120.55) | 615 (127.54)

2. Secondary Outcome: Nasal Secretion Weights
Description: Nasal secretions were collected in pre-weighed tissues and then weighed upon return for nasal secretion weight
Time Frame: each day for 5 days
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Number analyzed (Participants) | 11 | 22
grams
  Day 2 | 2.9 (0.618) | 0.8 (0.176)
  Day 3 | 2.0 (0.309) | 0.8 (0.276)
  Day 4 | 1.8 (0.420) | 0.8 (0.210)
  Day 5 | 2.0 (0.309) | 0.7 (0.276)
  Day 6 | 1.5 (0.301) | 0.8 (0.188)

3. Secondary Outcome: Severity of Symptom Scores - COUGH
Description: Cough symptoms were rated by the participant each day for 6 days and on day 30. Symptoms were rated from 0 - 3 corresponding to none, mild, moderate and severe, respectively.
Time Frame: once a day for six days and on day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Number analyzed (Participants) | 11 | 22
units on a scale
  Day 1 | 1.5 (0.121) | 0.7 (0.147)
  Day 2 | 1.6 (0.089) | 0.7 (0.145)
  Day 3 | 1.5 (0.121) | 0.7 (0.137)
  Day 4 | 1.3 (0.113) | 0.5 (0.118)
  Day 5 | 1.3 (0.071) | 0.4 (0.102)
  Day 6 | 0.7 (0.082) | 0.4 (0.104)
  Day 30 | 0.2 (0.071) | 0.1 (0.052)

4. Secondary Outcome: Severity of Symptom Score - NASAL CONGESTION
Description: nasal congestion symptoms were rated by the participant once a day for six days and on day 30. Symptoms were rated from 0 - 3 corresponding to none, mild, moderate and severe, respectively.
Time Frame: once a day for six days and on day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Number analyzed (Participants) | 11 | 22
units on a scale
  Day 1 | 1.5 (0.144) | 1.5 (0.14)
  Day 2 | 1.8 (0.106) | 1.4 (0.129)
  Day 3 | 1.7 (0.138) | 1.2 (0.139)
  Day 4 | 1.4 (0.118) | 1.0 (0.133)
  Day 5 | 1.3 (0.113) | 1.2 (0.117)
  Day 6 | 1.4 (0.118) | 1.1 (0.136)
  Day 30 | 0.4 (0.089) | 0.4 (0.104)

5. Secondary Outcome: Severity of Symptom Score - SNEEZING
Description: Sneezing symptoms were rated by participants once a day for six days and on Day 30, symptoms were rated from 0 - 3 corresponding to none, mild, moderate and severe, respectively.
Time Frame: once a day for six days and on Day 30
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Confirmed Respiratory Infection | Unconfirmed Respiratory Infection
Number analyzed (Participants) | 11 | 22
units on a scale
  Day 1 | 0.9 (0.095) | 0.9 (0.179)
  Day 2 | 0.9 (0.053) | 0.8 (0.179)
  Day 3 | 0.7 (0.113) | 0.7 (0.145)
  Day 4 | 0.7 (0.082) | 0.7 (0.145)
  Day 5 | 0.6 (0.089) | 0.6 (0.117)
  Day 6 | 0.5 (0.092) | 0.5 (0.14)
  Day 30 | 0.4 (0.089) | 0.2 (0.093)

ADVERSE EVENTS:
Arm/Group | Confirmed Respiratory Virus | Unconfirmed Respiratory Infection
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/22
Other Adverse Events (participants affected / at risk) | 0/11 | 0/22

LIMITATIONS AND CAVEATS:
Respiratory viruses were not detected in approximately 2/3 of the enrolled subjects. Future studies will need to apply more stringent inclusion/exclusion criteria to circumvent this problem.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes